CLINICAL TRIAL: NCT03465241
Title: Prospective, Open Clinical Study of Postoperative ctDNA Dynamic Monitoring and Its Role of Prognosis in Patients With Stage II to IIIA Non-small Cell Lung Cancer (NSCLC) Using Secondary Gene Sequencing (NGS)
Brief Title: ctDNA Dynamic Monitoring and Its Role of Prognosis in Stage II to IIIA NSCLC by NGS
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Other Study IDs: GASTO1035
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: NSCLC
Keywords: Non-Small Cell Lung Cancer; stage II to IIIA; circulating tumor DNA; The next generation of high-throughput gene sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, lymph node tissue, blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monitoring by NGS group: This group will accept the ctDNA dynamic monitoring on the following phase:the day before surgery,the 3rd to 7th day after surgery,3 to 4 weeks after adjuvant chemotherapy finished, then every 6 months in the following 2 years.
  Interventions: Diagnostic Test: the ctDNA dynamic monitoring

INTERVENTIONS:
Diagnostic Test: the ctDNA dynamic monitoring — To detect ctDNA in patients using the second generation of high-throughput gene sequencing (NGS)

SUMMARY:
The second generation of high-throughput gene sequencing (NGS) is an important means of detecting the tumor DNA and circulating tumor DNA (ctDNA), which can detect trace ctDNA from smaller plasma samples. This project is chiefly to study the role of ctDNA dynamic monitoring of stage IIA to IIIA NSCLC by NGS technique to verify the prognostic predictive effect of ctDNA. And the investigators also wander the concordance of lung cancer related genes mutation map and frequency between primary tumors and infiltrated regional lymph nodes.

DETAILED DESCRIPTION:
In the NGS era, ctDNA detection can truly reflect the real tumor tissue gene mutation map and frequency. It becomes the evaluation of therapeutic effect and the important monitoring indicators of clinical follow-up after surgery and adjuvant chemotherapy. The second generation of high-throughput gene sequencing (NGS) is an important means of detecting ctDNA, which can detect trace ctDNA from smaller plasma samples. The DNA dynamic monitoring of stage II to IIIA non-small cell lung cancer (NSCLC) was performed by the NGS technique to verify prognostic predictive effect of ctDNA in stage IIA to IIIA NSCLC patients after operation. The lung cancer related genes mutation map and frequency between primary tumors and infiltrated regional lymph nodes seems not exactly consistent. In this study, the investigators will compare the lung cancer related genes mutation map and frequency between primary tumors, bloodstream and infiltrated lymph node by the NGS technique.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative histopathological diagnosis of TNM stage IIA to IIIA NSCLC with R0 resection;
* No previous chemotherapy, radiotherapy, surgery or biological therapy for lung cancer；
* Eastern Cooperative Oncology Group (ECOG) behavior status score 0 to 1.

Exclusion Criteria:

* Patients with other cancers other than NSCLC within five years prior to this study;
* Who can not get enough tumor histological specimens (non-cytological) for analysis;
* Human immunodeficiency virus (HIV) infection;
* NSCLC mixed with patients with small cell lung cancer;
* Pregnant or lactating women;
* There is a clear history of neurological or mental disorders, including epilepsy or dementia;
* Conditions that investigators think is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Stage IIA to IIIA Non-small Cell Lung Cancer (NSCLC) with R0 resection.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years after the last patient enrolled
  Disease-free survival was assessed from surgery to disease recurrence or death as a result of any cause

SECONDARY OUTCOMES:
the genes mutation map and frequency between primary tumors, bloodstream and infiltrated lymph node | one month after the last patient enrolled
  we will compare the lung cancer related genes mutation map and frequency between primary tumors, bloodstream and infiltrated lymph node by the NGS technique.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li N, Wang BX, Li J, Shao Y, Li MT, Li JJ, Kuang PP, Liu Z, Sun TY, Wu HQ, Ou W, Wang SY. Perioperative circulating tumor DNA as a potential prognostic marker for operable stage I to IIIA non-small cell lung cancer. Cancer. 2022 Feb 15;128(4):708-718. doi: 10.1002/cncr.33985. Epub 2021 Oct 18. PMID 35076939